CLINICAL TRIAL: NCT05502939
Title: Effects of Music Training on Neurodevelopment and Associated Health Outcomes
Brief Title: Music Training and Child Development Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Assal Habibi, Associate Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UP-22-00056
Record Dates: First submitted 2022-08-10; First posted 2022-08-16 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Music
Keywords: Brain; Music training; Children

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Participants will not be masked to the intervention group assignment but will be blinded to the outcome measures.
  One research coordinator, fluent in English and in Spanish, will be unblinded to the participants' designated intervention. This individual will be responsible for all necessary follow up communications with the participants and their families.
  One graduate student research assistant will be unblinded to participant's designated intervention. They will be responsible for completing all fidelity and attendance measures. They will be in direct contact with program staff of the music and the afterschool enrichment program.
  Dr. Mack as the primary trial statistician and oversight on data analysis will be blinded to intervention assignments. All research staff involved in data analysis will be blinded to the intervention group assignment and all outcome measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Experimental): 57 participants, aged 6-8
  Participants will be enrolled in a music training program led by professional trained music instructor of the Colburn School of Music. The music curriculum follows the standard Suzuki training method. Students attend the program 3 days per week, 2 weekday afternoons and one weekend morning. Each session lasts approximately 1 hour long. Each student will be given a string instrument to take home (often a viola or a violin). Each learning day focuses on development of musical elements including rhythm and meter, form, pitch, and performance. Students will take part in annual performances intended to give them a motivational goal, sense of mastery and to share their accomplishments with their peers, family, and community.
  Interventions: Behavioral: Music Program
- After School Enrichment Group (Active Comparator): 57 participants, aged 6-8
  Participants will be enrolled in an after school program led by instructors and will include visual arts, theater, and general cultural studies. Students attend the program 3 days per week in the afternoon for 1 hour long lessons. Students will take part in an end of the year celebration to share their work with family and community members. Duration and frequency of the after-school program will be matched to the music intervention.
  Interventions: Behavioral: After School Enrichment Program

INTERVENTIONS:
Behavioral: Music Program — The cohort of students entering the program at the Colburn school in Los Angeles will be a part of a traditional strings curriculum. Students will join the program on a full scholarship and will be provided all materials necessary for instruction, including an instrument. Students will attend Colburn twice a week in a group setting and will receive private instruction once a week.
  The program will last 2, 15-week semesters (fall, spring) for 2-years. There will be 2 groups of 10 students. Students will undergo group instruction for 1 hour, 2 times a week and private instruction for 45 minutes, once a week.
  Arms: Music
Behavioral: After School Enrichment Program — The afterschool program will be led by instructors and will include visual arts, theater, and general cultural studies. Students attend the program 3 days per week in the afternoon for 1 hour long lessons. Students will take part in an end of the year celebration to share their work with family and community members.
  Arms: After School Enrichment Group

SUMMARY:
This proposed study aims to provide a definitive answer to whether music training benefits brain development, particularly brain inhibition control circuitry and its related health outcomes using a randomized control trial design.

In the study, 114 children between ages 6-8 from Los Angeles will be randomly assigned to a 24-month:(1) community-focused after school music training group focused on a traditional strings curriculum at the Colburn school in Los Angeles (MG) or (2) a control group (CG) after-school program comprising of visual arts, book club, ethnic and cultural studies and theater without specific focus on systematic music training or sports. Imaging data will be collected at before and after the intervention (24 months), behavioral assessments will be conducted before the intervention and yearly afterwards, and mid-intervention evaluations will be performed every six months throughout the study.

DETAILED DESCRIPTION:
The investigators will use an RCT design to investigate effects of a music training intervention on brain inhibition control circuitry. Throughout R61(N=40) and R33 (N=74) phases, 114 children between ages 6-8 from communities with limited resources in Los Angeles will be randomly assigned to a 24-month: (1) community-focused after school music training group focused on a traditional strings curriculum at the Colburn school in Los Angeles (MG) or (2) a control group (CG) after-school program comprising of visual arts, book club, ethnic and cultural studies and theater without specific focus on systematic music training or sports. Imaging data will be collected at before and after the intervention (24 months), behavioral assessments will be conducted before the intervention and yearly afterwards, and mid-intervention evaluations will be performed every six months throughout the study.

The investigators anticipate that the R61 phase will take 2 years and R33 will take 3 years to complete. The goal of the R61 phase is to evaluate the feasibility of executing the RCT. Comprehensive behavioral and imaging data will be collected at pre- and post-intervention, and mid-intervention evaluations will be performed every six months throughout the study. The combined R61/R33 phases will include 114 participants and will ultimately provide much needed guidance on the development of larger trials in the field.

ELIGIBILITY:
Inclusion Criteria:

* normal IQ (standard score of >85 in the Abbreviated Wechsler's Scale of Intelligence)
* Living in LA within 2 miles radius of the location of the music and the afterschool programs
* limited resources as defined by the Hollingshead Index cumulative score below 29
* ages 6-8

Exclusion Criteria:

* current diagnosis of neurological or psychiatric disorders
* prior engagement in formal and systematic music training for more than 6 months
* previous or current diagnosis of severe hearing loss defined as air conduction thresholds greater than 60 dB HL through 8 kHz or- severe vision loss that is not correctable with prescription eyeglasses or contact lenses
* non-removable, non-MRI compatible body parts
* Claustrophobia

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 114 (Estimated)
Dates: Start 2022-09-11 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
brain inhibition control networks | 24 months
  The primary outcome will be %change in blood-oxygen-level-dependent signal in the brain frontal circuits including the DLPFC, ACC and pre-SMA/SMA evaluated during the two inhibition control tasks.

SECONDARY OUTCOMES:
inhibition control as measured by reaction time | 24 months
  Stop signal reaction time during stop signal task
inhibition control as measured by delayed gratification | 24 months
  discounting rate from delay gratification task

CONTACTS AND LOCATIONS:
Overall Officials: Assal Habibi, Principal Investigator — University of Southern California
Locations (1):
- Brain and Creativity Institute, Los Angeles, California, United States